CLINICAL TRIAL: NCT06677320
Title: Establishing the Clinical Significance Values of Scales Used in Rotator Cuff Disease
Brief Title: Establishing Clinical Significance in Rotator Cuff Disease
Status: Recruiting | Type: Observational
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ozan Gür, PT, Research Assistant, Kırklareli University
Other Study IDs: 2024-1636
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Disease
Keywords: rotator cuff; clinical significance; minimal important chance; substantial clinical benefit; patient acceptable symptomatic state; maximal outcome improvement; Shoulder Disability Questionnaire; Western Ontario Rotator Cuff Index; Shoulder Rating Questionnaire; University of California-Los Angeles Shoulder Scale
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rotator cuff patients: Patients with rotator cuff disease who will receive conservative treatment.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Patients with rotator cuff disease will receive exercise treatment for two months.

SUMMARY:
The goal of this observational study is to learn about rotator cuff patients. The main questions it aims to answer are:

* What is the minimal clinically important difference value of the Shoulder Disability Questionnaire, the short version of the Western Ontario Rotator Cuff Index, the Shoulder Rating Questionnaire, and the University of California-Los Angeles Shoulder Scale?
* What is the substantial clinical benefit value of the Shoulder Disability Questionnaire, the short version of the Western Ontario Rotator Cuff Index, the Shoulder Rating Questionnaire, and the University of California-Los Angeles Shoulder Scale?
* What is the patient-acceptable symptomatic state value of the Shoulder Disability Questionnaire, the short version of the Western Ontario Rotator Cuff Index, the Shoulder Rating Questionnaire, and the University of California-Los Angeles Shoulder Scale?
* What is the maximal outcome improvement value of the Shoulder Disability Questionnaire, the short version of the Western Ontario Rotator Cuff Index, the Shoulder Rating Questionnaire, and the University of California-Los Angeles Shoulder Scale?
* What are the risk factors that prevent rotator cuff patients from reaching the minimal clinically important difference value?
* What are the risk factors that prevent rotator cuff patients from reaching the substantial clinical benefit value?
* What are the risk factors that prevent rotator cuff patients from reaching the patient-acceptable symptomatic state value?
* What are the risk factors that prevent rotator cuff patients from reaching the maximal outcome improvement value?

ELIGIBILITY:
Inclusion Criteria:

* to be over 18 years old
* to be a rotator cuff patient

Exclusion Criteria:

* to have another pathology in the affected shoulder area
* to have a neurological, rheumatological, or oncological disease
* to have radiculopathy
* to have had a previous fracture or operation in the affected shoulder area
* to be not cooperative enough for what will be done within the scope of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted with rotator cuff patients who will have physical therapy at Kırklareli Training and Research Hospital's physical therapy unit.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Functional level | before the treatment and within 1 week after 2 months of treatment
  Shoulder Disability Questionnaire (total score between 0-100) (higher values indicate higher disability)
Functional level | before the treatment and within 1 week after 2 months of treatment
  The short version of the Western Ontario Rotator Cuff Index (total score between 0-100) (higher values indicate higher functional level)
Functional level | before the treatment and within 1 week after 2 months of treatment
  Shoulder Rating Questionnaire (total score between 17-100) (higher values indicate higher functional level)
Functional level | before the treatment and within 1 week after 2 months of treatment
  The University of California-Los Angeles Shoulder Scale (total score between 0-100) (higher values indicate higher functional level)

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Gür, MSc, Principal Investigator — Kırklareli University
Locations (1):
- Kırklareli Eğitim ve Araştırma Hastanesi, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided